CLINICAL TRIAL: NCT05258032
Title: Structural and Functional Characterization of Rare Ocular Diseases
Acronym: RADIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Barcelona Macula Foundation (Other)
Responsible Party: Principal Investigator, Marc Biarnes Perez, PhD, Barcelona Macula Foundation
Other Study IDs: BarcelonaMaculaF
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Retinitis Pigmentosa; Stargardt Disease 1; Best Disease; Pattern Dystrophy of Macula; Choroideremia
Keywords: Retinitis pigmentosa; Stargardt's disease 1; Best disease; Pattern Dystrophy of Macula; Choroideremia
MeSH Terms: conditions — Retinitis Pigmentosa; Stargardt Disease; Vitelliform Macular Dystrophy; Choroideremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rare ocular diseases (ROD) are a heterogeneous group of ocular diseases that affect very few people and, generally, for which no tretament is available. An important subgroup of these diseases are inherited retinal degenerations. In this study we focus on understanding the natural history of different ROD that affect the posterior segment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older with a diagnosis of a ROD affecting the posterior segment
* Patients able to undergo all required ophthalmic exams
* Patients able and willing to sign an informed consent

Exclusion Criteria:

* Patients with other concomitant posterior segment disorders
* Patients taking drugs known to affect the retina and/or optic nerve
* Patients that underwent an intraocular surgery (aside from phacoemulsification with intraocular lens implantation), corneal or glaucoma surgery
* Patients who have participated in the past 12 months or that are currently participating in clinical trials for an ocular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a ROD affecting the posterior segment of the eye
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-11-24 (Estimated); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Change in best corrected visual acuity | Year 2 as compared to baseline
  Change from baseline in BCVA

SECONDARY OUTCOMES:
Change in mean macular sensitivity | Year 2 as compared to baseline
  Change from baseline in mean macular sensitivity on microperimetry
Change in retinal thickness | Year 2 as compared to baseline
  Change from baseline in central subfield retinal thickness on OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de la màcula, Barcelona, Spain